CLINICAL TRIAL: NCT06562049
Title: Carpal Bone Erosion in Rheumatoid Arthritis :Diagnostic Value
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abeer Abdelaal Aly, resident of Physical medicine, Rheumatology and Rehabilitation Department, Sohag University
Other Study IDs: soh-med-24-07-10MS
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cases: rheumatoid arthriris patients
  Interventions: Radiation: musculoskeletal ultrasound
- control: systemic lupus patients
  Interventions: Radiation: musculoskeletal ultrasound
- controls: healthy controls
  Interventions: Radiation: musculoskeletal ultrasound

INTERVENTIONS:
Radiation: musculoskeletal ultrasound — musculoskeletal ultrasound on both hands

SUMMARY:
Rheumatoid arthritis (RA) is a systemic inflammatory disease characterized by proliferative hyper vascularized synovitis which primarily affects synovial joints. Synovium of bursa; tendon sheaths; attachment sites of cartilage, ligament, and tendons to the bone; soft tissue; and bones can be mentioned among the other areas under influence of RA. Changes happen to be symmetrical and may present as fusiform soft tissue swelling, regional osteoporosis, marginal-central erosions, cartilage damage, joint destruction, narrowing of joint space and fibrous ankyloses. Wrist, metacarpophalangeal and metatarsophalangeal joints are the first sites to be affected .Over the past few years, an increasing number of rheumatologists have started to use US in the clinical setting of the early arthritis clinic. While US allows for an accurate and non-invasive multisite assessment of joint involvement in patients with RA, time for US examination is not infinite

ELIGIBILITY:
Inclusion Criteria:

* 1. RA patients fulfilled the 2010 American College of Rheumatoid Arthritis classification criteria.[8] 2. SLE patients fulfilled the 2019 ACR\EULAR classification criteria for SLE.[9] 3. Age above 18 years old. 4. Patient cooperative and can answer questions. 5. Patients who are able and willing to give written informed consent.

Exclusion Criteria:

* 1. Age below 18 years and above 60 years. 2. Uncooperative patients. 3. Patient not able and willing to give written informed consent.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. RA patients fulfilled the 2010 American College of Rheumatoid Arthritis classification criteria.[8]
  2. SLE patients fulfilled the 2019 ACR\EULAR classification criteria for SLE.[9]
  3. Age above 18 years old.
  4. Patient cooperative and can answer questions.
  5. Patients who are able and willing to give written informed consent
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
bone erosion | max 1 year
  erosions in carpal bones and MCP 2,5 in both hands

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sommer OJ, Kladosek A, Weiler V, Czembirek H, Boeck M, Stiskal M. Rheumatoid arthritis: a practical guide to state-of-the-art imaging, image interpretation, and clinical implications. Radiographics. 2005 Mar-Apr;25(2):381-98. doi: 10.1148/rg.252045111. PMID 15798057
- [Background] Ejbjerg BJ, Vestergaard A, Jacobsen S, Thomsen H, Ostergaard M. Conventional radiography requires a MRI-estimated bone volume loss of 20% to 30% to allow certain detection of bone erosions in rheumatoid arthritis metacarpophalangeal joints. Arthritis Res Ther. 2006;8(3):R59. doi: 10.1186/ar1919. Epub 2006 Mar 15. PMID 16542505
- [Background] Mottonen TT. Prediction of erosiveness and rate of development of new erosions in early rheumatoid arthritis. Ann Rheum Dis. 1988 Aug;47(8):648-53. doi: 10.1136/ard.47.8.648. PMID 3137902